CLINICAL TRIAL: NCT00531986
Title: HIV- Monotherapy in Switzerland (MOST- ch)
Brief Title: HIV - Monotherapy in Switzerland (MOST-ch)
Acronym: MOST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unexpectedely high rates of treatment-failure
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: Swiss National Science Foundation (Other); Swiss HIV Cohort Study (Network)
Responsible Party: Principal Investigator, pietro vernazza, Director Division Infectious Diseases, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHCS-Projekt Nr.: 490; SHCS 490
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: HIV Infections
Keywords: Monotherapy; Neuropsychological tests; HIV viral load in ZNS; HIV viral load in genital; Lumbar puncture and HIV viral load in ZNS; Monotherapy and compartment failure (ZNS and genital); ZNS viral load under monotherapy; Genital viral load under monotherapy; Neuropsychological tests (HIV Dementia); Treatment Experienced
MeSH Terms: conditions — HIV Infections; AIDS Dementia Complex | interventions — lopinavir-ritonavir drug combination; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monotherapy (Experimental): Ritonavir-boosted lopinavir (Kaletra®) will be used as monotherapy
  Interventions: Drug: Lopinavir-Monotherapy
- Continued ART (Active Comparator): Continuation Therapy, conventional triple HAART
  Interventions: Drug: HAART

INTERVENTIONS:
Drug: Lopinavir-Monotherapy — Patients on triple HAART will be switched to LPV/r-monotherapy
  Other Names: Kaletra
  Arms: Monotherapy
Drug: HAART — Patients will continued their current HAART
  Other Names: Any ART
  Arms: Continued ART

SUMMARY:
The investigators plan to conduct a two arm study, to compare failure rates in the central nervous system (CNS) and genital compartment in virologically fully suppressed patients continuing a highly active antiretroviral therapy (HAART) versus patients switching to ritonavir boosted lopinavir (Kaletra®) HIV-monotherapy. The study is composed of two phases of 48 weeks duration.

In addition, neuropsychological tests (Color trial test A 1 and 2; Grooved pegboard; EWIA Digit Symbol form) and evaluation of side effects will be performed.

DETAILED DESCRIPTION:
In the first phase (phase A), ritonavir-boosted lopinavir (Kaletra®) will be compared with continued HAART. In the second year (phase B) patients on conventional HAART are also offered LPV/r monotherapy to extend the longterm experience of this new strategy.

Only patients willing to give a genital secretion and a spinal fluid sample will be included. All patients must be on a fully suppressive HAART with at least 2 consecutive values of HIV-RNA at the screening visit . After performance of lumbar puncture at baseline, patients will be randomized to continued HAART or LPV/r monotherapy. During the first year of randomized treatment patients will be followed at week 6/ 12 /18 /24 /32 /40 and 48. Lumbar puncture and genital secretion sampling will be repeated at week 48.

Follow up during the second phase (B: W48-96) of the study will be identical to phase A including genital and spinal sampling at week 96. After study termination at week 96, patients may opt to continue monotherapy if results of HIV-RNA in blood and CSF support this decision.

The primary endpoint of the study will be treatment failure in the compartment (CSF and / or genital tract). Since the variability of HIV-RNA determination in CSF and genital secretions is not very well known, a one log increase above the baseline value will be considered as treatment failure in the respective compartment. Only patients who had a complete viral suppression in blood will be considered for compartment evaluation. Patients treated in the monotherapy arm with a CSF HIV-RNA value at week 48 more than 1.0 log10 cp/ml above baseline (= compartment failure) will be switched to a conventional combination treatment. HIV-RNA testing in the genital samples will be performed batchwise at the end of the study.

In addition, patients with a blood treatment failure (two consecutive HIV-RNA detections > 400cp/ml) will be considered as full treatment failures and switched to a rescue regimen at the discretion of the treating physician. For the analysis, these patients will be considered as systemic treatment failure and will not be entered in the analysis of compartmentalized treatment failure. If the rescue strategy was only intensification of adherence and results in full blood viral load re-suppression, the patient will still be maintained in the study and compartment evaluations can be performed at w48 and/or 96, respectively.

The secondary aim of the study is the definition of prognostic markers for compartment failures. Potential risk factors associated with mono-maintenance failure are HIV-DNA load at time of treatment simplification, HIV-RNA at the time of first treatment initiation, duration of HIV-RNA suppression before simplification, history of HIV-RNA blips, presence of detectable HIV-RNA in spinal fluid at the time of treatment simplification, changes of level of c-reactive protein (high sensitive methodology, hsCRP) from baseline as a marker of immune-activation during the maintenance therapy.

If funding allows, we will test for the presence of resistant viruses and compare the presence of genetic polymorphism at baseline. We will also measure parameters of immunoactivation (hsCRP, CD8+, CD38+).

The study is financed by the Swiss National Science Foundation and the Swiss HIV Cohort Study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* HIV seropositive.
* HAART (> 6 months) with at least 3 months successfully suppressed HIV- RNA (two most recent RNA measurements < 50 cp/ml). HAART is defined as either:

  * 1 PI plus 2 NRTIs,
  * 1 NNRTI plus 2 NRTIs, or
  * 3 NRTIs.
* HIV-RNA in plasma < 50 cp/ml at screening.
* Stable antiretroviral therapy (unchanged drug combination) during the last four weeks.
* If not currently on a LPV/ r based therapy, willing to switch to LPV/ r bid therapy in case patient is randomized to the monotherapy arm
* Signed written informed consent.
* Highly motivated patients able to understand the investigational nature of this open observational study and willing to participate in additional procedures.

Exclusion Criteria:

* Other investigational substance or substances active against HIV.
* Previous history of adverse events with the drugs under investigation.
* Previous history of any virological treatment failure (does not include deliberate treatment interruption) or documented resistance against the drugs under investigation (LPV/r).
* Patient who has no effective alternative treatment options in case the study treatment fails (according to the physician's judgment).
* Pregnancy (negative pregnancy test for women of childbearing potential at screening).
* Active AIDS-defining disease necessitating antibiotic or chemotherapy at the time of screening.
* Chronic hepatitis B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Failure in CNS | Week 48

SECONDARY OUTCOMES:
Predictors of failure | week 48

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Vernazza, Professor, Principal Investigator — Swiss HIV Cohort Study
Locations (6):
- Switzerland (6):
  - Flepp, Zurich, Bellariastrasse 38
  - Furrer, Bern, INF KP PKT 2B Freiburgstr.
  - Nuesch, Basel, Petersgraben 4
  - Cavassini, Lausanne, Rue Du Bugnon 21
  - Opravil, Zurich, Rämistrasse 100
  - Hirschel, Geneva

REFERENCES:
- [Derived] Gutmann C, Cusini A, Gunthard HF, Fux C, Hirschel B, Decosterd LA, Cavassini M, Yerly S, Vernazza PL; Swiss HIV Cohort Study (SHCS). Randomized controlled study demonstrating failure of LPV/r monotherapy in HIV: the role of compartment and CD4-nadir. AIDS. 2010 Sep 24;24(15):2347-54. doi: 10.1097/QAD.0b013e32833db9a1. PMID 20802298
- See also: Related Info — http://www.infekt.ch